CLINICAL TRIAL: NCT05869825
Title: High Flow Nasal Cannula and Non-Invasive Positive Pressure Ventilation Following Extubation in Infants After Cardiac Surgery for Congenital Heart Disease: A Randomized Clinical Trial
Brief Title: HFNC vs NIPPV Following Extubation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Asaad Beshish, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003745
Record Dates: First submitted 2023-03-30; First posted 2023-05-22 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Congenital Heart Disease
Keywords: Cardiac surgery for CHD; Cardiac Intensive Care Unit
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The high-flow nasal cannula (HFNC) (Active Comparator): The high flow nasal cannula (HFNC) is a unique mode of respiratory support that delivers warmed, humidified oxygen with a wide range of fractions of inspired oxygen (FiO2) and flow rate (liters/min) without an invasive device such as an endotracheal tube (breathing tube).
  Interventions: Procedure: High Flow Nasal Canula following extubation
- Non-invasive positive pressure ventilation (NIPPV) (Active Comparator): Non-invasive positive pressure ventilation (NPPV or NIPPV) is a unique mode of respiratory support that delivers pressurized, oxygen-enriched gas to the airway via the nose and/or oropharynx without a more invasive device such as an endotracheal tube (breathing tube).
  Interventions: Procedure: Non-Invasive Positive Pressure Ventilation following extubation

INTERVENTIONS:
Procedure: High Flow Nasal Canula following extubation — Participants in this group will be randomized to receive High Flow Nasal Cannula support after extubation. The patient will be clinically monitored and respiratory support will be escalated per a specific flow sheet. The patient will remain on this assigned air support method until they are either removed entirely from air support or need to be re-intubated with oxygen.
  Other Names: HFNC
  Arms: The high-flow nasal cannula (HFNC)
Procedure: Non-Invasive Positive Pressure Ventilation following extubation — Participants in this group will be randomized to receive NIPPV respiratory support following extubation. The patient will be clinically monitored and respiratory support will be escalated per a specific flow sheet. The patient will remain on this assigned air support method until they are either removed entirely from air support or need to be re-intubated with oxygen.
  Other Names: NIPPV
  Arms: Non-invasive positive pressure ventilation (NIPPV)

SUMMARY:
This study has the goal to determine the best method of respiratory support following extubation after cardiac surgery (CS). After cardiac surgery for Congenital Heart Disease (CHD), patients remain intubated until the cardiac team determines it is safe for the patient to undergo a trial of extubation. Two common methods of respiratory support following extubation are High Flow Nasal Cannula (HFNC) and Non Invasive Positive Pressure Ventilation (NIPPV). There is currently a gap in data comparing High Flow Nasal Cannula and Non-Invasive Positive Pressure Ventilation in infants (age 0-1) in regard to extubation failure and overall outcomes.

This study will monitor the health outcomes of 200 infants (0 - 1 year) with CHD following cardiac surgery in the Cardiac Intensive Care Unit (CICU) at Children's Healthcare of Atlanta (CHOA). This will be done by assigning the respiratory support method each child will receive following extubation after cardiac surgery. Health outcomes will be monitored until discharge or until the second instance of extubation failure.

Both study arms are standard-of-care respiratory support methods in the CHOA CICU. The investigators aim to determine which of these two methods has fewer risk factors when used with infants.

DETAILED DESCRIPTION:
This study aims to answer an important clinical question that all providers struggle with: how to optimize respiratory support following extubation in Infants After Cardiac Surgery (CS) for Congenital Heart Disease (CHD). The high morbidity and at times mortality associated with failed extubation events demonstrates this clearly, as extubation failure (EF) is stressful to this fragile population and results in hemodynamic compromise as well as airway trauma due to manipulation of the airway.

This study aims to: 1) comparatively examine which mode of respiratory support (HFNC vs NIPPV) after extubation is more effective at lowering rates of EF, and 2) examine clinical risk factors, outside of the respiratory support model (HFNC vs. NIPPV), that are associated with EF in patients with CHD after CS.

These infants often remain endotracheally intubated on mechanical ventilatory support upon return to the Cardiac Intensive Care Unit (CICU). These patients undergo a trial of extubation at the discretion of the CICU team when deemed safe. Studies have shown that approximately 3-27% of patients with CHD fail extubation after cardiac surgery. Risk factors for extubation failure (EF) are complex surgical repair, younger age, smaller patients, presence of airway anomalies, genetic abnormalities, pulmonary hypertension, use of cardiopulmonary bypass (CPB), hypothermia, atelectasis, lung injury, phrenic and diaphragmatic nerve injury, and prolonged open sternotomy. Patients with CHD who are successfully extubated using NIPPV have been shown to have shorter lengths of stay, while studies in pre-term infants without CHD showed NIPPV reduced EF compared to hood/tent oxygen, or HFNC. Other studies have shown HFNC to decrease the need for intubation in infants with respiratory failure and may improve respiratory mechanics through unidirectional flow in the upper airway, decreasing dead space, improving minute ventilation, pulmonary compliance, and distending airway pressure. This support ultimately reduces the work of breathing and oxygen consumption, while enhancing oxygen delivery.

Despite the use of HFNC and NIPPV to support patients following extubation, there is limited data on the comparative effectiveness of HFNC versus NIPPV to prevent EF in infants with CHD after CS. The investigators hypothesize that the use of HFNC will be associated with lower rates of EF, and a shorter length of stay when compared to NIPPV.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the CICU following cardiac surgery for CHD who are </= 1 year of age and/or weight </= 10 kg

Exclusion Criteria:

* Patients who remain intubated for >/= 4 weeks
* Patients who have a tracheostomy in place prior to their cardiac surgery
* Patient enrolled in a competing research study
* Patients requiring extracorporeal membrane oxygenation (ECMO) support preoperatively
* Patients with birth weight < 2 Kg.
* Gestational age < 35 weeks at birth.
* Patients with extracardiac anomalies more than minor severity.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To compare the effectiveness in avoiding extubation failures of High Flow Nasal Cannula (HFNC) vs Non-Invasive Positive Pressure Ventilation (NIPPV) | After surgery up to 2 weeks
  Rates of extubation failures (EF) will be compared among both groups. Data will be collected from the hospital electronic medical record system.

SECONDARY OUTCOMES:
Patient's clinical breathing status at discharge | At hospital discharge up to a year
  The research team will review the hospital's electronic medical record and check the patient's breathing status (oxygen saturation on room air) after the patient's hospital discharge
Difference of patients' clinical hemodynamical status at discharge | At hospital discharge up to a year
  The research team will review the hospital's electronic medical record and check the patient's vital signs (blood pressure and heart rate) to determine the clinical hemodynamical status at discharge.
Length of hospital stay difference between treatment groups | From hospital admission until hospital discharge up to a year
  The research team will review the hospital's electronic medical records after the patient's hospital discharge. The length of hospital stay (days) will be calculated from time of hospital admission until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Asaad Beshish, MD, Principal Investigator — Emory University
Locations (1):
- Arthur M. Blank Hospital | Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The research team will present the analyzed data at conferences and will also be submitted for publication.